CLINICAL TRIAL: NCT03698383
Title: Phase II Study of Trastuzumab Biosimilar (Herzuma®) Plus Gedatolisib in Patients With HER-2 Positive Metastatic Breast Cancer Who Progressed After 2 or More HER-2 Directed Chemotherapy
Brief Title: Phase II Study of Herzuma® Plus Gedatolisib in Patients With HER-2 Positive Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Kyong-Hwa, Park, Professor, Korean Cancer Study Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG-BR18-13/TR-03
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: HER2-positive Breast Cancer; Metastatic Breast Cancer
Keywords: Herzuma; Gedatolisib
MeSH Terms: conditions — Breast Neoplasms | interventions — gedatolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Herzuma plus Gedatolisib (Experimental)
  Interventions: Drug: Trastuzumab biosimilars(Herzuma), Gedatolisib

INTERVENTIONS:
Drug: Trastuzumab biosimilars(Herzuma), Gedatolisib — * Trastuzumab biosimilar: Intravenously administered on Day 1 of every 21 day cycle at a dose of 6mg/kg (loading dose 8mg/kg at 1C)
  * Gedatolisib: Intravenously administered on Day 1, 8 and 15 of every 21 day cycle at a dose of 180mg
  Other Names: Herzuma plus Gedatolisib

SUMMARY:
Phase II Pilot Study of Trastuzumab Biosimilar (Herzuma®) plus Gedatolisib in Patients with HER-2 Positive Metastatic Breast Cancer Who Progressed after 2 or more HER-2 directed Chemotherapy

DETAILED DESCRIPTION:
All the patients will be included in the final analysis, with a total of 15 patients to be enrolled.

Treatment will occur until disease progression, unacceptable toxicity or patient withdrawal.

Tumor measurement and evaluation are going to be performed at every 6 weeks for the first 3 months, then at every 9 weeks till progression, and then follow-up evaluation at every 12 weeks thereafter end of study.

ELIGIBILITY:
Inclusion Criteria:

* Breast tumor with suspected PI3K-pathway dependence (either by mutation or by known biologic rationale. PI3K dependence includes the presence of a PIK3CA-mutant hotspot mutation, PIK3CA copy number gain, mTOR hotspot mutation, or PTEN loss in the archival or fresh tumor tissue specimen identified in K-MASTER panel. All genetic findings must be reviewed by the study PI, prior to study entry.).
* Patient is an adult, female ≥ 19 years old at the time of informed consent.
* Patient has histologically and/or cytologically confirmed diagnosis of HER2-positive breast cancer. HER2-positive breast cancer as defined by an immunohistochemistry (IHC) score of 3+ or gene amplified by in situ hybridization (ISH) as defined by a ratio of ≥ 2.0 for the number of HER2 gene copies to the number of chromosome 17 copies.Metastatic or unresectable disease documented on diagnostic imaging studies.
* Metastatic or unresectable disease documented on diagnostic imaging studies.
* Prior 2 or more HER-2 directed therapy including trastuzumab for metastatic disease is mandatory.
* Patient must have at least one measurable lesion according to Response valuation Criteria in Solid Tumors version 1.1 (RECIST v.1.1).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
* Adequate bone marrow and organ function including: WBC ≥ 3500/mL; Platelets ≥ 100,000/uL; Hemoglobin >9.0 g/dL; Total bilirubin ≤ 1.5x ULN; AST and ALT < 2.5 x ULN; Alkaline phosphatase <2.5x ULN; Creatinine ≤ 1.5x ULN or CCr >60 ml/min for patients with abnormal serum Cr level function.
* Adequate glucose control, as defined by HbA1c < 7% and fasting blood glucose ≤ 126 mg/dL (7.0 mmoL/L).
* Adequate glucose control, as defined by HbA1c < 7% and fasting blood glucose ≤ 126 mg/dL (7.0 mmoL/L).
* Life expectancy higher than 3 months
* Patient has an adequate left ventricular ejection function of at least 50 % at baseline, as measured by echocardiography.
* Written informed consent

Exclusion Criteria:

* Patient is pregnant or lactating, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
* Patient has received previous treatment with a mechanistic target of rapamycin (mTOR) inhibitor or phosphoinositide 3-kinase (PI3K) inhibitor.
* Patient has symptomatic and unstable CNS metastases, except for treated brain metastases. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed.
* Active and clinically significant bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus syndrome (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness. Baseline viral assessment is not required in patients with no known infection.
* Current use or anticipated need for food or medications that are known moderate or greater CYP3A4 inhibitors, including their administration within 7-days prior to the first gedatolisib dose and while receiving investigational product (ie, strong CYP3A4 inhibitors: grapefruit juice or grapefruit/grapefruit related citrus fruits [e.g., Seville oranges, pomelos], ketoconazole, miconazole, itraconazole, voriconazole, posaconazole, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, amprenavir, fosamprenavir nefazodone, lopinavir, troleandomycin, mibefradil, conivaptan; moderate CYP3A4 inhibitors: erythromycin, verapamil, atazanavir, delavirdine, fluconazole, darunavir, diltiazem, aprepitant, imatinib, tofisopam, ciprofloxacin, and cimetidine).
* Concurrent use or anticipated need for medications that are mainly metabolized by UGT1A9 including their administration within 7-days prior to the first dose of investigational product (e.g., propofol, propranolol, dapagliflozin, darexaban, mycophenolic acid, and tapentadol).
* Acetaminophen use within 24 hours before or after the first dose of gedatolisib.
* Current use or anticipated need for food or medications that are metabolized by CYP2D6, and of narrow therapeutic index including their administration within 10-days prior to the first gedatolisib dose and while receiving investigational product.
* Concurrent use of herbal preparations.
* Major surgery within 4 weeks of first dose of investigational product or not fully recovered from any side effects of previous procedures.
* Any other malignancy within 3 years prior to first dose of investigational product except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
* QTc interval >480 msec (based on the mean value of the triplicate ECGs), family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation or Torsade de Pointes.
* Any of the following within 6 months of first dose of investigational product myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of NCI CTCAE v. 5.0 Grade ≤2, atrial fibrillation of any grade, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident including transient ischemic attack, or symptomatic pulmonary embolism.
* History of interstitial pneumonitis.
* Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | within maximum 3 years
  the percentage of patients experiencing confirmed complete response (CR) and partial response (PR) assessed by RECIST criteria v.1.1

SECONDARY OUTCOMES:
Progression free survival | within maximum 3 years
  the time from study entry until the first observation of disease progression according to the above schedule or death due to any cause
Overall survival | within maximum 3 years
  the time from study entry until death

CONTACTS AND LOCATIONS:
Overall Officials: Kyong Hwa Park, MD, PhD, Principal Investigator — Korean Cancer Study Group
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harbeck N, Huang CS, Hurvitz S, Yeh DC, Shao Z, Im SA, Jung KH, Shen K, Ro J, Jassem J, Zhang Q, Im YH, Wojtukiewicz M, Sun Q, Chen SC, Goeldner RG, Uttenreuther-Fischer M, Xu B, Piccart-Gebhart M; LUX-Breast 1 study group. Afatinib plus vinorelbine versus trastuzumab plus vinorelbine in patients with HER2-overexpressing metastatic breast cancer who had progressed on one previous trastuzumab treatment (LUX-Breast 1): an open-label, randomised, phase 3 trial. Lancet Oncol. 2016 Mar;17(3):357-366. doi: 10.1016/S1470-2045(15)00540-9. Epub 2016 Jan 26. PMID 26822398
- [Background] Wong HH, Collins J, McAdam K, Wilson C. Trastuzumab beyond progression in advanced breast cancer: national guidance versus oncologist's decision. Oncology. 2014;86(1):22-3. doi: 10.1159/000356876. Epub 2013 Dec 10. No abstract available. PMID 24335099
- [Background] Rexer BN, Arteaga CL. Optimal targeting of HER2-PI3K signaling in breast cancer: mechanistic insights and clinical implications. Cancer Res. 2013 Jul 1;73(13):3817-20. doi: 10.1158/0008-5472.CAN-13-0687. Epub 2013 Jun 21. PMID 23794708
- [Background] Wang L, Yu X, Wang C, Pan S, Liang B, Zhang Y, Chong X, Meng Y, Dong J, Zhao Y, Yang Y, Wang H, Gao J, Wei H, Zhao J, Wang H, Hu C, Xiao W, Li B. The anti-ErbB2 antibody H2-18 and the pan-PI3K inhibitor GDC-0941 effectively inhibit trastuzumab-resistant ErbB2-overexpressing breast cancer. Oncotarget. 2017 May 16;8(32):52877-52888. doi: 10.18632/oncotarget.17907. eCollection 2017 Aug 8. PMID 28881779
- [Background] Courtney KD, Corcoran RB, Engelman JA. The PI3K pathway as drug target in human cancer. J Clin Oncol. 2010 Feb 20;28(6):1075-83. doi: 10.1200/JCO.2009.25.3641. Epub 2010 Jan 19. PMID 20085938
- [Background] Del Campo JM, Birrer M, Davis C, Fujiwara K, Gollerkeri A, Gore M, Houk B, Lau S, Poveda A, Gonzalez-Martin A, Muller C, Muro K, Pierce K, Suzuki M, Vermette J, Oza A. A randomized phase II non-comparative study of PF-04691502 and gedatolisib (PF-05212384) in patients with recurrent endometrial cancer. Gynecol Oncol. 2016 Jul;142(1):62-69. doi: 10.1016/j.ygyno.2016.04.019. Epub 2016 Apr 24. PMID 27103175
- [Background] Janku F, Wheler JJ, Naing A, Falchook GS, Hong DS, Stepanek VM, Fu S, Piha-Paul SA, Lee JJ, Luthra R, Tsimberidou AM, Kurzrock R. PIK3CA mutation H1047R is associated with response to PI3K/AKT/mTOR signaling pathway inhibitors in early-phase clinical trials. Cancer Res. 2013 Jan 1;73(1):276-84. doi: 10.1158/0008-5472.CAN-12-1726. Epub 2012 Oct 12. PMID 23066039
- [Background] Baselga J, Cortes J, Im SA, Clark E, Ross G, Kiermaier A, Swain SM. Biomarker analyses in CLEOPATRA: a phase III, placebo-controlled study of pertuzumab in human epidermal growth factor receptor 2-positive, first-line metastatic breast cancer. J Clin Oncol. 2014 Nov 20;32(33):3753-61. doi: 10.1200/JCO.2013.54.5384. Epub 2014 Oct 20. PMID 25332247
- [Background] Hurvitz SA, Andre F, Jiang Z, Shao Z, Mano MS, Neciosup SP, Tseng LM, Zhang Q, Shen K, Liu D, Dreosti LM, Burris HA, Toi M, Buyse ME, Cabaribere D, Lindsay MA, Rao S, Pacaud LB, Taran T, Slamon D. Combination of everolimus with trastuzumab plus paclitaxel as first-line treatment for patients with HER2-positive advanced breast cancer (BOLERO-1): a phase 3, randomised, double-blind, multicentre trial. Lancet Oncol. 2015 Jul;16(7):816-29. doi: 10.1016/S1470-2045(15)00051-0. Epub 2015 Jun 16. PMID 26092818
- [Background] Andre F, Hurvitz S, Fasolo A, Tseng LM, Jerusalem G, Wilks S, O'Regan R, Isaacs C, Toi M, Burris H, He W, Robinson D, Riester M, Taran T, Chen D, Slamon D. Molecular Alterations and Everolimus Efficacy in Human Epidermal Growth Factor Receptor 2-Overexpressing Metastatic Breast Cancers: Combined Exploratory Biomarker Analysis From BOLERO-1 and BOLERO-3. J Clin Oncol. 2016 Jun 20;34(18):2115-24. doi: 10.1200/JCO.2015.63.9161. Epub 2016 Apr 18. PMID 27091708
- [Background] Mauro C, Smith J, Cucchi D, Coe D, Fu H, Bonacina F, Baragetti A, Cermenati G, Caruso D, Mitro N, Catapano AL, Ammirati E, Longhi MP, Okkenhaug K, Norata GD, Marelli-Berg FM. Obesity-Induced Metabolic Stress Leads to Biased Effector Memory CD4+ T Cell Differentiation via PI3K p110delta-Akt-Mediated Signals. Cell Metab. 2017 Mar 7;25(3):593-609. doi: 10.1016/j.cmet.2017.01.008. Epub 2017 Feb 9. PMID 28190771
- [Background] Roychoudhuri R, Eil RL, Restifo NP. The interplay of effector and regulatory T cells in cancer. Curr Opin Immunol. 2015 Apr;33:101-11. doi: 10.1016/j.coi.2015.02.003. Epub 2015 Feb 27. PMID 25728990
- [Background] Patton DT, Wilson MD, Rowan WC, Soond DR, Okkenhaug K. The PI3K p110delta regulates expression of CD38 on regulatory T cells. PLoS One. 2011 Mar 1;6(3):e17359. doi: 10.1371/journal.pone.0017359. PMID 21390257
- [Background] Pearce VQ, Bouabe H, MacQueen AR, Carbonaro V, Okkenhaug K. PI3Kdelta Regulates the Magnitude of CD8+ T Cell Responses after Challenge with Listeria monocytogenes. J Immunol. 2015 Oct 1;195(7):3206-17. doi: 10.4049/jimmunol.1501227. Epub 2015 Aug 26. PMID 26311905
- [Background] Crompton JG, Sukumar M, Roychoudhuri R, Clever D, Gros A, Eil RL, Tran E, Hanada K, Yu Z, Palmer DC, Kerkar SP, Michalek RD, Upham T, Leonardi A, Acquavella N, Wang E, Marincola FM, Gattinoni L, Muranski P, Sundrud MS, Klebanoff CA, Rosenberg SA, Fearon DT, Restifo NP. Akt inhibition enhances expansion of potent tumor-specific lymphocytes with memory cell characteristics. Cancer Res. 2015 Jan 15;75(2):296-305. doi: 10.1158/0008-5472.CAN-14-2277. Epub 2014 Nov 28. PMID 25432172
- [Background] Marshall NA, Galvin KC, Corcoran AM, Boon L, Higgs R, Mills KH. Immunotherapy with PI3K inhibitor and Toll-like receptor agonist induces IFN-gamma+IL-17+ polyfunctional T cells that mediate rejection of murine tumors. Cancer Res. 2012 Feb 1;72(3):581-91. doi: 10.1158/0008-5472.CAN-11-0307. Epub 2011 Dec 9. PMID 22158905
- [Background] Muraro E, Comaro E, Talamini R, Turchet E, Miolo G, Scalone S, Militello L, Lombardi D, Spazzapan S, Perin T, Massarut S, Crivellari D, Dolcetti R, Martorelli D. Improved Natural Killer cell activity and retained anti-tumor CD8(+) T cell responses contribute to the induction of a pathological complete response in HER2-positive breast cancer patients undergoing neoadjuvant chemotherapy. J Transl Med. 2015 Jun 27;13:204. doi: 10.1186/s12967-015-0567-0. PMID 26116238
- [Background] Shapiro GI, Bell-McGuinn KM, Molina JR, Bendell J, Spicer J, Kwak EL, Pandya SS, Millham R, Borzillo G, Pierce KJ, Han L, Houk BE, Gallo JD, Alsina M, Brana I, Tabernero J. First-in-Human Study of PF-05212384 (PKI-587), a Small-Molecule, Intravenous, Dual Inhibitor of PI3K and mTOR in Patients with Advanced Cancer. Clin Cancer Res. 2015 Apr 15;21(8):1888-95. doi: 10.1158/1078-0432.CCR-14-1306. Epub 2015 Feb 4. PMID 25652454
- [Background] Fruman DA, Meyers RE, Cantley LC. Phosphoinositide kinases. Annu Rev Biochem. 1998;67:481-507. doi: 10.1146/annurev.biochem.67.1.481. PMID 9759495